CLINICAL TRIAL: NCT06933888
Title: Assessment of Nutritional Knowledge, Habits, and Eating Behavior in Athletic Women to Evaluate the Possible Impact on Their Menstrual Function
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Rossella Nappi, Principal investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: P_6620
Record Dates: First submitted 2025-03-27; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Hypothalamic Amenorrhea, Functional
Keywords: Functional Hypothalamic Amenorrhea; Eating disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The present study aims to investigate the degree of knowledge about nutrition and dietary habits in athletic women through validated questionnaires and to evaluate a possible impact on their menstrual function, including women with a diagnosis of functional hypothalamic amenorrhea (FHA) and women who present with a different menstrual dysfunction (oligomenorrhea or polymenorrhea in absence of organic causes).

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 16-30 years
* Physical activity > 2 days per week
* Informed consent from the patient and/or an authorized legal representative

Exclusion Criteria:

* Menstrual disorders of organic cause (ovarian cysts, uterine fibroids, polyps, etc.)
* Concomitant non-reproductive organic diseases (hypertension, diabetes, etc.)
* Use of psychopharmacological therapies
* Language barrier

Ages: 16 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: Young athletic women referred for menstrual dysfunction of non-organic causes
Sampling Method: Non-Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Assess nutritional knowledge in athletic women with functional hypothalamic amenorrhea | Baseline
  The outcome will be assessed with a single measurement through a validated questionnaire (General and Sport Nutrition Knowledge [GeSNK]). More specifically, the proportion of subjects with moderate knowledge (score between 46 and 58) will be evaluated.

SECONDARY OUTCOMES:
Evaluation of nutritional knowledge in athletic women with menstrual dysfunctions of different nature, comparing women with FHA to those with oligomenorrhea/polymentorrhea in the absence of organic diseases. | Baseline
  Assessment of nutritional knowledge through GeSNK questionnaire in women with menstrual dysfunction of non-organic cause other than functional hypothalamic amenorrhea
Assessment of eating habits in in athletic women with menstrual dysfunctions of different nature, comparing women with FHA to those with oligomenorrhea/polymentorrhea in the absence of organic diseases | Baseline
  Assessment of eating habits and nutritional intake through a food diary to identify the presence of low energy availability.
Evaluation of eating behavior in athletic women with menstrual dysfunctions of different nature, comparing women with FHA to those with oligomenorrhea/polymentorrhea in the absence of organic diseases. | Baseline
  Assessment of Low Energy Availability in Females questionnaire [LEAF-Q]
Evaluation of eating behavior in athletic women with menstrual dysfunctions of different nature, comparing women with FHA to those with oligomenorrhea/polymentorrhea in the absence of organic diseases. | Baseline
  Assessment of Eating Attitude Test 26 [EAT-26]
Evaluation of eating behavior in athletic women with menstrual dysfunctions of different nature, comparing women with FHA to those with oligomenorrhea/polymentorrhea in the absence of organic diseases. | Baseline
  Assessment of Eating Disorder Inventory -2 [EDI-2]
Evaluation of eating behavior in athletic women with menstrual dysfunctions of different nature, comparing women with FHA to those with oligomenorrhea/polymentorrhea in the absence of organic diseases. | Baseline
  Assessment of ORTO-15 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SSD Ostetricia e Ginecologia 2 - Riproduzione e Procreazione Medicalmente Assistita, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No